CLINICAL TRIAL: NCT04525391
Title: Phase II, Single-arm Study of AZD2811 and Durvalumab (MEDI4736) Combination Therapy in Relapsed Small Cell Lung Cancer Subjects [SUKSES-N5]
Brief Title: AZD2811 and Durvalumab (MEDI4736) Combination Therapy in Relapsed Small Cell Lung Cancer
Acronym: SUKSES-N5
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recommended completion of the study due to SUSAR occurring in other clinical trials conducted with the same drug.
Sponsor: Se-Hoon Lee (Other)
Responsible Party: Sponsor-Investigator, Se-Hoon Lee, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUKSES-N5
Record Dates: First submitted 2020-08-14; First posted 2020-08-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: SCLC, Recurrent
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab+AZD2811 to SCLC patients (Experimental): Dosage and Schedule: AZD2811 500mg and durvalumab 1500mg via IV administered on Day 1 for every 3weeks (fixed dosing for subjects > 30 kg body weight for durvalumab). One cycle is consisted of 3 weeks.
  The drug products must be dosed consecutively using different infusion lines. The sequence of infusions is as follows: durvalumab is administered first over 1 hour, followed by AZD2811 administered over 2 hours. A waiting time interval of at least 30 minutes between the end of durvalumab infusion and start of AZD2811 infusion should be adhered to.
  Interventions: Drug: Durvalumab+AZD2811 to SCLC patients

INTERVENTIONS:
Drug: Durvalumab+AZD2811 to SCLC patients — AZD2811 must NOT be infused through a 0.2-µm or 0.22-µm filter and therefore durvalumab and AZD2811 MUST be infused through different infusion lines. In order not to exceed the endotoxin limit, durvalumab and AZD2811 mustbe administered consecutively. Durvalumab is administered first over 1 hour, followed by AZD2811 administered over 2 hours. AZD2811 should be administered at 30 minutes after the end of the durvalumab infusion, as long as there are no acute infusion reactions to durvalumab.

SUMMARY:
Samsung Medical Centre, Seoul, Korea. Additional 0~5 Korea Lung Cancer Consortium (KLCC) centres in Korea Up to 40 subjects will be enrolled in two-stages (first stage: 19 evaluable subjects and second stage: 17 evaluable subjects and additional 4 subjects considering the drop out rate) If the study is conducted as de-escalated dosage (Durvalumab 1120mg) after the safety run-in, number of the patients will be counted from the second safety-run in phase.

DETAILED DESCRIPTION:
This study is a single arm, open-label, multi-centre phase II study of AZD2811NP and durvalumab combination therapy in subjects with relapsed small cell lung cancer (SCLC) as a second or third line treatment.

Subjects will receive AZD2811 and durvalumab combination therapy. The arm is composed of up to approximately 36 evaluable subjects.

After the initiation of the study, a safety run-in period will be conducted with 6 patients to confirm the safety profile.

Thus a safety run-in will be undertaken in the first 6 patients with 1500mg of Durvalumab q 3weeks with 500mg of AZD2811. During the safety follow-up, if 2 or more DLT is observed, another safety run-in with new 6 patients will be initiated with 1120mg of Durvalumab q 3weeks with 500mg of AZD2811.

In case of a positive risk benefit profile the recruitment will continue.

Subjects will receive AZD2811 500mg and durvalumab 1500mg via IV administered on Day 1 for every 3weeks (fixed dosing for subjects > 30 kg body weight). One cycle consists of 3 weeks. The sequence of the infusion is Durvalumab administered over 1 hour, followed by AZD2811 administered over 2 hours. The optimal proposed time between infusions is 15 min to 30 min. The compatibility of drug products in infusion line has not been tested. Therefore, the infusion line must be flushed with saline after the administration of one drug product and before the start of the second drug product.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Subjects must be ≥ 18 years of age.
3. Body weight > 30kg
4. Small cell lung cancer that has progressed during or after first-line therapy.

   1. The 1st line regimen must have contained platinum based regimen and must have documented radiological and/or clinical progression on treatment.
   2. Refractory to first-line chemotherapy or relapse within 6 months since the last dose of first-line chemotherapy
   3. If the subject has sensitive relapse (relapse more than 6 months since the last dose of first-line chemotherapy), (s)he should receive second-line treatment prior to study entry.
5. Histologically confirmed SCLC with documented c-MYC expression (≥ c-MYC IHC 1+)
6. Subjects are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
7. ECOG performance status 0-1
8. Subjects must have a life expectancy ≥ 3months from proposed first dose date.
9. Subjects must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

   1. Haemoglobin ≥ 9.0g/dL)
   2. White blood cells (WBC) ≥ 3 x 109/L
   3. Platelet count ≥ 100 x 109/L
   4. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   5. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
   6. Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN
   7. Subjects must have serum creatinine (CR) ≤1.5 times the normal upper limit of the study institution or creatinine clearance estimated using the Cockcroft-Gault equation of ≥ 45 mL/min: Estimated creatinine clearance = (140-age [years]) x weight (kg) (x F)a serum creatinine (mg/dL) x 72 a where F=0.85 for females and F=1 for males.
10. At least one measurable lesion that can be accurately assessed at baseline by imaging or physical examination at baseline and is suitable for repeated assessment.
11. Postmenopausal or evidence of non-childbearing status for women of childbearing Potential or a negative urine or serum pregnancy test at screening and confirmed prior to treatment on Day 1 of every cycle

    Postmenopausal is defined as:
    1. Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
    2. Luteinizing hormone(LH) and Follicle stimulating hormone(FSH) levels in the post menopausal range for women under 50
    3. Radiation-induced oophorectomy with last menses >1 year ago
    4. Chemotherapy-induced menopause with >1 year interval since last menses
    5. Surgical sterilisation(bilateral oophorectomy or hysterectomy)
12. Male and women of childbearing portential , who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination, throughout the period of taking study treatment and for 6 months after last dose of investigational product(s) to prevent pregnancy in a partner.
13. Provision of tumor sample (from either archival and/or fresh biopsy)
14. Optional: Provision of separate informed consent for genetic research. If a subject declines to participate in the genetic research, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this Clinical Study Protocol, so long as they consent to the main informed consent.

Exclusion Criteria:

1. Previous enrolment in the present study or concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
2. More than two prior chemotherapy regimens for the treatment of small cell lung cancer refractory to first-line chemotherapy or relapse within 6 months.

   (However, immunotherapy is not counted the prior chemotherapy regimen.)
3. Subjects with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for > 2 years. Or patients with a history of leptomeningeal carcinomatosis.
4. Treatment with any investigational product during the last 14 days before the first dose on study.
5. Subjects receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The subject can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment.
6. Receiving, or having received, concomitant medications, herbal supplements and/or foods that significantly modulate cytochrome P450 3A4(CYP3A4) or P-glycoprotein(P-gp) activity (washout periods of 2 weeks, but 3 weeks for St. John's Wort). Note these include common azole antifungals, macrolide antibiotics and other medications.
7. Prior exposure to an AURKB inhibitor or PD-1 or PD-L1 or CTLA-4 inhibitor.
8. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

   1. Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection)
   2. Systemic corticosteroids at physiologic doses not to exceed 10mg/day of prednisone or its equivalent
   3. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
9. Receipt of live attenuated vaccine within 30 days prior to the first dose of investigational product. Note: Subjects, if enrolled, should not receive live vaccine whilst receiving investigational product and up to 180 days after the last dose of investigational product.
10. Any unresolved toxicity NCI CTCAE grade≥2 from previous anticancer therapy with the exception of alopecia, vitilgo, and the laboratory values defined in the inclusion criteria (CTCAE version 5.0)

    1. Subjects with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Investigator.
    2. Subjects with irreversible toxicity not reasonably expected to be exacerabated by treatment with durvalumab may be included only after consultation with with the Investigator.
11. Intestinal obstruction or CTCAE grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.
12. Haematuria: +++ on microscopy or dipstick
13. INR ≥ 1.5 or other evidence of impaired hepatic synthesis function
14. Subject has any of the following cardiac criteria:

    1. Mean QT interval corrected for heart rate(QTcF) ≥ 470ms calculated from 3 electrocardiograms (ECGs) using Fridericia's correction.
    2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, third degree heart block, second degree heart block, first degree heart block.
    3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40years of age or any concomitant medication known to prolong the QT interval.
    4. Uncontrolled hypertension-blood pressure (BP) ≥ 150/95mmHg despite medical therapy.
    5. Unstable atrial fibrillation or unstable cardiac arrhythmia with a ventricular rate > 100bpm on an ECG at rest.
    6. Symptomatic heart failure - New York Heart Association Grade II to Grade IV.
    7. Prior or current cardiomyopathy.
    8. Severe valvular heart disease.
    9. Uncontrolled angina (Canadian Cardiovascular Society Grade II to Grade IV despite medical therapy) or acute coronary syndrome within 6months prior to screening.
    10. Subjects at risk of brain perfusion problems (e.g., carotid stenosis hypotension, including a fall in blood pressure of > 20mm Hg)
15. Female subjects who are pregnant or breast-feeding or child-bearing or male or female subjects of reproductive potential who are not willing to employ effective birth control from screening to 6 months after the last dose of durvalumab or AZD2811.
16. Any evidence of severe or uncontrolled intercurrent illness, including but limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the subject to give written informed consent.
17. History of allogenic organ transplantation.
18. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), Hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Subjects with a past or resolved HBV infection (defined as the antibody[anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
19. Known hypersensitivity to any of the study drugs or any of the study drug excipients.
20. Known central nervous system (CNS) disease other than neurologically stable, treated brain metastases - defined as metastasis having no evidence of progression or haemorrhage for at least 2 weeks after treatment.
21. Major surgical procedures ≤ 28 days of beginning study treatment, or minor (outpatient) surgical procedures ≤ 7days
22. History of active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease, diverticulitis [with the exception of diverticulosis], systemic lupus erythematosis, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]).

The following are exceptions to this criterion:

1. Subjects with vitiligo or alopecia
2. Subjects with hypothyroidism(e.g., following Hashimoto syndrome) stable on hormone replacement
3. Any chronic skin condition that dose not require systemic therapy
4. Subjects without active disease in the last 5 years may be included but only after consultation with the Investigator.
5. Subjects with cardiac disease controlled by diet alone

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Disease control rate is defined as the proportion of patients with best response of CR, PR, or who have SD for at least 12 weeks | 12 weeks
  To investigate the efficacy of AZD2811 and durvalumab combination therapy in subjects with relapsed SCLC subjects with c-MYC expression ≥ 1+ as 2nd or 3rd line therapy

SECONDARY OUTCOMES:
Duration of response (SD, PR, CR) calculated by Kaplan-Meier method | 12 weeks
  To assess secondary measures of clinical efficacy
Overall survival(OS) calculated by Kaplan-Meier method | 12 weeks
  To assess secondary measures of clinical efficacy
Progression-free survival(PFS) calculated by Kaplan-Meier method | 12 weeks
  To assess secondary measures of clinical efficacy
Time to first relapse (resistant relapse or sensitive relapse) | 12 weeks
  Planned subgroup analyses

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided